CLINICAL TRIAL: NCT01722604
Title: Therapeutic Equivalence Study of Generic Brinzolamide vs Azopt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CD-11-265
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2021-06

CONDITIONS: Glaucoma; Open Angle or Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — brinzolamide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azopt 1% ophthalmic suspension (Active Comparator): Ophthalmic suspension
  Interventions: Drug: Azopt 1%
- Brinzolamide 1% ophthalmic suspension (Experimental): ophthalmic suspension
  Interventions: Drug: brinzolamide 1% ophthalmic suspension

INTERVENTIONS:
Drug: brinzolamide 1% ophthalmic suspension — brinzolamide 1% ophthalmic suspension
  Arms: Brinzolamide 1% ophthalmic suspension
Drug: Azopt 1% — Azopt 1%, RLD
  Arms: Azopt 1% ophthalmic suspension

SUMMARY:
The main purpose of this prospective study is to demonstrate the therapeutic equivalence of topical brinzolamide dosed three times daily compared with AzoptTM (brinzolamide ophthalmic suspension 1%) dosed three times daily in IOP reduction in patients with POAG or OH.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years of age or older,
* diagnosed with primary open-angle glaucoma or ocular hypertension.

Exclusion Criteria:

* Patients with any form of glaucoma (such as secondary, congenital, juvenile or normal tension glaucoma, angle closure glaucoma) in either eye other than primary open-angle glaucoma,
* ocular hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- US01, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
Started | 129 | 129
Completed | 123 | 120
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Full Range); unit: years] | 64.1 [39 to 91] | 65.3 [39 to 89] | 64.6 [39 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 81 | 159
  Male | 51 | 48 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 32 | 61
  White | 97 | 97 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Week 12
Time Frame: Week 12
Population: The Per Protocol (PP) Population was utilized for the primary outcome. All randomized participants who completed both the baseline visit (eligibility visit 2) and the week 12 visit and who had no major protocol violations, and who also completed week 4 and week 8 visits, were included in the PP population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
Number analyzed (Participants) | 122 | 124
mmHg | 20.6 (3.21) | 20.8 (3.37)

2. Secondary Outcome: Change in Intraocular Pressure (IOP) From Baseline to Week 12
Time Frame: Baseline, Week 12
Population: The Per Protocol (PP) Population was utilized for the secondary outcome. All randomized participants who completed both the baseline visit (eligibility visit 2) and the week 12 visit and who had no major protocol violations, and who also completed week 4 and week 8 visits, were included in the PP population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
Number analyzed (Participants) | 122 | 124
mmHg | -5.3 (2.79) | -5.4 (3.27)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 2/129 | 3/129
Other Adverse Events (participants affected / at risk) | 9/129 | 5/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinzolamide 1% Ophthalmic Suspension (N=129) | Azopt 1% Ophthalmic Suspension (N=129)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinzolamide 1% Ophthalmic Suspension (N=129) | Azopt 1% Ophthalmic Suspension (N=129)
Instillation site complication (General disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.